CLINICAL TRIAL: NCT01691950
Title: Investigating the Outcomes of Lower-limb Trauma Patients
Brief Title: Investigating Outcomes of Lower Limb Trauma
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Engineering and Physical Sciences Research Council, UK (Other)
Responsible Party: Sponsor
Other Study IDs: CRO1934
Record Dates: First submitted 2012-04-23; First posted 2012-09-25 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Trauma
Keywords: Trauma; Limb reconstruction; Amputation; Functional outcome; Sensing
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reconstruction: Those who have undergone limb reconstruction following lower limb trauma
- Healthy volunteers: Healthy volunteers for control

SUMMARY:
This is an observational study, which aims to firstly develop a sensor-based objective mobility assessment. This will then be used to profile and compare the outcomes of patients who undergo amputation with those who have limb salvage surgery following a traumatic injury to their lower limb.

DETAILED DESCRIPTION:
In the setting of severe trauma, the decision whether to amputate or save a limb is common, and extremely difficult to make. Due to improving reconstructive surgical techniques there are currently no clear criteria for amputation. Although limb salvage appears desirable in most situations, numerous articles in the scientific literature have shown that it is associated with increased pain, complications, duration of hospital stay, rehabilitation time, and overall costs. These factors may be acceptable if the patients benefited from improved functional outcome. However, studies comparing amputation to limb salvage consistently report no significant difference in functional outcome between the two groups.

A major limitation in the methodology of the fore mentioned studies is the use of self-reported questionnaires to determine functional outcome. Questionnaires are subjective, and often lack specificity, and therefore may not be truly representative of functional outcome. Furthermore, lack of useful information during long-term post-operative care prevents adaption and optimisation of rehabilitation strategies.

The investigators plan on using a wearable sensor to develop an objective mobility assessment tool for patients having either amputation or limb salvage surgery after lower limb trauma. This would result in a reliable and accurate comparison, which may help healthcare professionals make an informed decision between amputation and limb salvage in the future.

ELIGIBILITY:
Inclusion Criteria:

* To have sustained a lower-limb trauma and undergone limb salvage surgery OR amputation with fitting of prosthesis

Exclusion Criteria:

1. Contralateral (or other) limb impairment
2. 18 > AGE > 65
3. Currently a hospital inpatient
4. Psychological disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who have been treated following lower limb trauma at the Imperial College NHS Trust sites will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Kwasnicki, BSc (Hons), Principal Investigator — Imperial College London; Shehan Hettiaratchy, PhD, FRCS, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Healthy volunteers
Period: Overall Study
Arm/Group | Reconstruction | Control
Started | 20 | 10
Completed | 10 | 10
Not Completed | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reconstruction | Control | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (15.8) | 34.7 (12.9) | 36.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 18 | 9 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcome (Consisting of Questionnaire Score, Hamlyn Mobility Score (HMS) Gait/Activities of Daily Living Parameters)
Description: The Hamlyn Mobility Score is a measure of functional mobility as measured by a wearable sensors during simple physical activities. The score range is from 0 - 60, with 60 being the best score possible and represents normal physical function of a healthy adult.
Time Frame: 3 months post-reconstruction
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reconstruction | Control
Number analyzed (Participants) | 20 | 10
units on a scale | 19.7 (13.9) | 58.2 (1.6)

2. Secondary Outcome: Participant Length of Hospital Stay
Description: These measurements refer to the participants healthcare journey (which are not affected by the research project). Hospital stay refers to the time around their lower limb trauma and any further admissions.
Time Frame: Up to length of study (1-2 years)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Reconstruction | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10

LIMITATIONS AND CAVEATS:
The trial recruited 0 patients with prostheses and as such this study arm has been deleted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes